CLINICAL TRIAL: NCT00903383
Title: A Phase 2, Multi-center, Randomized, Double Blind, Placebo-controlled, Multiple-dose Study to Determine the Safety and Efficacy of Daily Orally Administered LX3305 in Subjects With Active Rheumatoid Arthritis (RA) on Stable Methotrexate (MTX) Therapy
Brief Title: Study of LX3305 in Subjects With Active Rheumatoid Arthritis on Stable Methotrexate
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Lexicon Pharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: Protocol LX3305.1-201-RA; LX3305.201, LX2931
Record Dates: First submitted 2009-05-14; First posted 2009-05-18 (Estimated); Results first posted 2011-12-15 (Estimated); Last update posted 2011-12-15 (Estimated); Status verified 2011-11

CONDITIONS: Rheumatoid Arthritis
MeSH Terms: conditions — Arthritis, Rheumatoid

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (4):
- Low Dose (Experimental): A low dose of LX3305; daily oral intake for 12 weeks
  Interventions: Drug: LX3305 low dose
- Mid Dose (Experimental): A mid dose of LX3305; daily oral intake for 12 weeks
  Interventions: Drug: LX3305 mid dose
- High Dose (Experimental): A high dose of LX3305; daily oral intake for 12 weeks
  Interventions: Drug: LX3305 high dose
- Placebo (Placebo Comparator): Matching placebo dosing with daily oral intake for 12 weeks
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: LX3305 low dose — A low dose of LX3305; daily oral intake for 12 weeks
  Arms: Low Dose
Drug: LX3305 mid dose — A mid dose of LX3305; daily oral intake for 12 weeks
  Arms: Mid Dose
Drug: LX3305 high dose — A high dose of LX3305; daily oral intake for 12 weeks
  Arms: High Dose
Drug: Placebo — Matching placebo dosing with daily oral intake for 12 weeks
  Arms: Placebo

SUMMARY:
The purpose of the study is to evaluate the safety, tolerability, and effectiveness of LX3305 versus a placebo control in subjects with active rheumatoid arthritis on stable methotrexate therapy.

ELIGIBILITY:
Inclusion Criteria:

* Males and females aged 18-75 years old
* Rheumatoid arthritis present for at least 6 months, functional class I, II, or III as defined by ACR criteria
* Active disease as determined by the presence of ≥6 swollen joints, ≥6 tender joints, and serum C-reactive protein level > upper limit of normal
* Receiving stable dose of MTX (≥10 mg/wk) and folate supplementation at least 8 weeks prior to Day 1
* Ability to provide written informed consent

Exclusion Criteria:

* RA diagnosis prior to 16 years of age (Juvenile RA)
* Lack of response to >3 disease modifying anti-rheumatic drugs (DMARDs) or exposure to >1 biologic DMARD
* Use of DMARDs other than MTX within 12 weeks prior to Day 1
* Intra-articular and/or parenteral corticosteroids within 4 weeks prior to study Day 1
* Blood donation or receipt of live vaccine within 4 weeks prior to Day 1
* Major surgical procedure within 8 weeks prior to Day 1
* Any systemic inflammatory condition, recurrent infection, or current infection other than onychomycosis
* History of cancer within 5 years prior to Day 1
* Presence of hepatic or biliary disease
* History of tuberculosis
* History of human immunodeficiency virus (HIV)

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 208 (Actual)
Dates: Start 2009-07; Primary Completion 2010-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Joel P. Freiman, MD, MPH, Study Director — Lexicon Pharmaceuticals, Inc.
Locations (38):
- United States (13):
  - Lexicon Investigational Site, Gainesville, Florida
  - Lexicon Investigational Site, Orange Park, Florida
  - Lexicon Investigational Site, Orlando, Florida
  - Lexicon Investigational Site, Tampa, Florida
  - Lexicon Investigational Site, Cumberland, Maryland
  - Lexicon Investigational Site, Hagerstown, Maryland
  - Lexicon Investigational Site, Kalamazoo, Michigan
  - Lexicon Investigational Site, Flowood, Mississippi
  - Lexicon Investigational Site, Hickory, North Carolina
  - Lexicon Investigational Site, Philadelphia, Pennsylvania
  - Lexicon Investigational Site, Nashville, Tennessee
  - Lexicon Investigational Site, Dallas, Texas
  - Lexicon Investigational Site, La Crosse, Wisconsin
- Bulgaria (5):
  - Lexicon Investigational Site, Pleven
  - Lexicon Investigational Site, Plovdiv
  - Lexicon Investigational Site, Rousse
  - Lexicon Investigational Site, Sofia
  - Lexicon Investigational Site, Veliko Tarnovo
- Czechia (4):
  - Lexicon Investigational Site, Bruntál
  - Lexicon Investigational Site, Hlučín
  - Lexicon Investigational Site, Sokolov
  - Lexicon Investigational Site, Zlín
- Hungary (6):
  - Lexicon Investigational Site, Békéscsaba
  - Lexicon Investigational Site, Budapest
  - Lexicon Investigational Site, Kecskemét
  - Lexicon Investigational Site, Makó
  - Lexicon Investigational Site, Sopron
  - Lexicon Investigational Site, Veszprém
- Poland (8):
  - Lexicon Investigational Site, Bialystok
  - Lexicon Investigational Site, Działdowo
  - Lexicon Investigational Site, Gdynia
  - Lexicon Investigational Site, Katowice
  - Lexicon Investigational Site, Lublin
  - Lexicon Investigational Site, Warsaw
  - Lexicon Investigational Site, Wroclaw
  - Lexicon Investigational Site, Włoszczowa
- Serbia (2):
  - Lexicon Investigational Site, Belgrade
  - Lexicon Investigational Site, Niška Banja

RESULTS

PARTICIPANT FLOW:
Recruitment Details: There were 43 study centers in 6 countries (10 in the US, 8 in Bulgaria, 4 in Czech Republic, 7 in Hungary, 11 in Poland, and 3 in Serbia). The first subject was enrolled on 31 August 2009, and the last subject completed the study on 30 September 2010.
Pre-assignment Details: There was a 4 week screening period prior to the 12-week treatment period.
Period: Overall Study
Arm/Group | Low Dose | Mid Dose | High Dose | Placebo
Started | 55 | 54 | 50 | 49
Completed | 48 | 48 | 47 | 44
Not Completed | 7 | 6 | 3 | 5
Not completed — Adverse Event | 1 | 2 | 3 | 1
Not completed — Physician Decision | 1 | 2 | 0 | 0
Not completed — Lost to Follow-up | 0 | 0 | 0 | 1
Not completed — Decision of Sponsor | 1 | 0 | 0 | 0
Not completed — Withdrawal by Subject | 4 | 1 | 0 | 2
Not completed — Patient Decision - Lack of Efficacy | 0 | 1 | 0 | 0
Not completed — Patient Decision | 0 | 0 | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Low Dose | Mid Dose | High Dose | Placebo | Total
Number analyzed (Participants) | 55 | 54 | 50 | 49 | 208
Age Continuous [Mean (Standard Deviation); unit: years] | 56.5 (9.25) | 55.8 (9.20) | 56.4 (10.89) | 57.5 (10.19) | 56.5 (9.83)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 47 | 43 | 37 | 41 | 168
  Male | 8 | 11 | 13 | 8 | 40

OUTCOME MEASURES:

1. Primary Outcome: ACR20 Response at Week 12
Description: Evaluates the efficacy of LX3305 by utilizing the American College of Rheumatology 20% response criteria (ACR20) at 12 weeks in subjects with active RA also receiving stable doses of MTX. For a response of ACR20, there had to be ≥20% improvement in swollen joint count, ≥20% improvement in painful/tender joint count, and ≥20% improvement in at least 3 of the following: subject's assessment of pain, global assessment of disease activity, assessment of physical function, or acute phase reactant (C-reactive protein or erythrocyte sedimentation rate).
Time Frame: Baseline and 12 weeks
Population: Intent to Treat Population
Measure: Number; unit: Participants
Arm/Group | Low Dose | Mid Dose | High Dose | Placebo
Number analyzed (Participants) | 55 | 54 | 50 | 49
Participants | 24 | 22 | 30 | 24

2. Secondary Outcome: ACR50 Response at Week 12
Description: Evaluates the efficacy of LX3305 by utilizing the American College of Rheumatology 50% response criteria (ACR50) at 12 weeks in subjects with active RA also receiving stable doses of MTX. For a response of ACR50, there had to be ≥50% improvement in swollen joint count, ≥50% improvement in painful/tender joint count, and ≥50% improvement in at least 3 of the following: subject's assessment of pain, global assessment of disease activity, assessment of physical function, or acute phase reactant (C-reactive protein or erythrocyte sedimentation rate).
Time Frame: Baseline and 12 weeks
Population: Intent to Treat Population
Measure: Number; unit: Participants
Arm/Group | Low Dose | Mid Dose | High Dose | Placebo
Number analyzed (Participants) | 55 | 54 | 50 | 49
Participants | 6 | 5 | 11 | 12

3. Secondary Outcome: ACR70 Response at Week 12
Description: Evaluates the efficacy of LX3305 by utilizing the American College of Rheumatology 70% response criteria (ACR70) at 12 weeks in subjects with active RA also receiving stable doses of MTX. For a response of ACR70, there had to be ≥70% improvement in swollen joint count, ≥70% improvement in painful/tender joint count, and ≥70% improvement in at least 3 of the following: subject's assessment of pain, global assessment of disease activity, assessment of physical function, or acute phase reactant (C-reactive protein or erythrocyte sedimentation rate).
Time Frame: Baseline and 12 weeks
Population: Intent to Treat Population
Measure: Number; unit: Participants
Arm/Group | Low Dose | Mid Dose | High Dose | Placebo
Number analyzed (Participants) | 55 | 54 | 50 | 49
Participants | 2 | 4 | 5 | 3

4. Secondary Outcome: Hybrid ACR Response at Week 12
Description: Evaluates the improvement in active RA by combining elements of the ACR20/50/70 with a continuous score of the mean change in core set measures. The percentage improvement from baseline was computed in each of the components of the ACR. The average percent improvement was calculated and used with the subject's ACR20, ACR50, and ACR70 status to compute the hybrid ACR response, with a positive change indicating improvement.
Time Frame: Baseline and 12 weeks
Population: Intent to Treat Population
Measure: Mean (Standard Deviation); unit: Percent change
Arm/Group | Low Dose | Mid Dose | High Dose | Placebo
Number analyzed (Participants) | 55 | 54 | 50 | 49
Percent change | 26.595 (23.2280) | 27.422 (24.3453) | 37.356 (26.1357) | 35.290 (24.4368)

5. Secondary Outcome: Change From Baseline in C-reactive Protein (mg/L) at Week 12
Description: The C-reactive protein value (mg/L) at baseline was subtracted from the value for each of the treatment groups at Week 12.
Time Frame: Baseline and 12 weeks
Population: Intent to Treat Population
Measure: Mean (Standard Deviation); unit: mg/L
Arm/Group | Low Dose | Mid Dose | High Dose | Placebo
Number analyzed (Participants) | 55 | 54 | 50 | 49
mg/L | -0.026 (15.7225) [-1.5071 to 17.4208] | 5.342 (26.5937) [2.0924 to 24.5573] | -5.316 (19.1959) [-7.3324 to 12.6649] | -7.983 (28.5387) [0 to 0]

6. Secondary Outcome: Change From Baseline in Erythrocyte Sedimentation Rate (mm) at Week 12
Description: The value for Erythrocyte Sedimentation Rate (mm) at baseline was subtracted from the value for each of the treatment groups at Week 12.
Time Frame: Baseline and 12 weeks
Population: Intent to Treat Population
Measure: Mean (Standard Deviation); unit: mm
Arm/Group | Low Dose | Mid Dose | High Dose | Placebo
Number analyzed (Participants) | 55 | 54 | 50 | 49
mm | -2.5 (21.23) [-3.00 to 13.18] | -3.3 (20.23) [-3.59 to 12.07] | -9.7 (21.76) [-10.32 to 6.17] | -7.6 (18.05) [0 to 0]

ADVERSE EVENTS:
Time Frame: Adverse events were followed during the 12-week Treatment period and during the 30-day Follow-up period.
Arm/Group | Low Dose | Mid Dose | High Dose | Placebo
Serious Adverse Events (participants affected / at risk) | 2/55 | 0/54 | 0/50 | 0/49
Other Adverse Events (participants affected / at risk) | 10/55 | 5/54 | 10/50 | 12/49
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Low Dose (N=55) | Mid Dose (N=54) | High Dose (N=50) | Placebo (N=49)
Nausea and Vomiting (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Atrial Fibrillation (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Low Dose (N=55) | Mid Dose (N=54) | High Dose (N=50) | Placebo (N=49)
Urinary Tract Infection (Infections and infestations) | 3 (4) | 1 (1) | 3 (5) | 6 (6)
Diarrhea (Gastrointestinal disorders) | 2 (2) | 3 (3) | 2 (3) | 1 (1)
Rheumatoid Arthritis (Musculoskeletal and connective tissue disorders) | 2 (2) | 1 (1) | 3 (3) | 2 (2)
Headache (Nervous system disorders) | 3 (3) | 0 (0) | 2 (2) | 3 (3)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The sponsor requires that written permission be given before the PI can release any data publicly.